CLINICAL TRIAL: NCT06065826
Title: Correlation Between Forward Head Posture And Myogenic Temporomandibular Disorder In Addicted Smartphone Users
Brief Title: Forward Head Posture and Myogenic TMD Association in Smartphone Overuse
Status: Completed | Type: Observational
Sponsor: Doha Hany Mohamed Labib (Other)
Responsible Party: Sponsor-Investigator, Doha Hany Mohamed Labib, Assistant lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: FHP and MTMD in SMP
Record Dates: First submitted 2023-08-29; First posted 2023-10-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Temporomandibular Disorder
Keywords: forward head posture; smartphone
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects with myogenic TMD: Subjects diagnosed as myogenic TMD according to the presence of trigger points in masseter, temporalis, upper trapezius and C5-C6 articular pillars Subjects are heavy smartphones users, using the SAS-SV, the cuffof value for males is 31 and for females is 33.
  Subjects have forward head posture assessed by CVA <49.9 degrees
  Interventions: Other: Assessment
- subjects without myogenic TMD: Subjects are heavy smartphones users, using the SAS-SV, the cuffof value for males is 31 and for females is 33.
  Subjects have forward head posture assessed by CVA <49.9 degrees
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — All subjects will be assessed for FHP by taking a lateral view picture to calculate the CVA using the Kinovea software. Each subject with FHP will be examined for myofascial trigger points done by the therapist finger to palpate bilaterally on tender nodules in masticatory and neck muscles. Then using a pressure algometer, the PPT value will be scored for each trigger in each muscle bilaterally. Masticatory muscle endurance will be measured by asking the subject to bite on load sensor for as long as the subject can until exhaustion. Using a stopwatch, the time will be recorded in seconds. Using the craniocervical extension endurance test, the subject will lie prone with their head unsupported and with a bubble inclinometer attached to their head. Using a stopwatch, time in seconds will be recorded to test how long the subject can sustain the neck in neutral position. Finally, a smartphone addiction scale will be answered by the subject to identify how much they are addicted to its use.

SUMMARY:
The goal of this observational study is to determine the correlation between forward head posture and myogenic temporomandibular disorder, pain pressure threshold and endurance of masticatory and neck muscles in addicted smart phone users. The main question it aims to answer is:

• What is the correlation between forward head posture and myogenic temporomandibular disorder, pain pressure threshold and endurance of masticatory and neck muscles in addicted smart phone users?

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) and cervical spine are closely related to each other due to their anatomical, mechanical and neurophysiological relationships. That's why pain and dysfunction in the cervical spine can be observed in patients with temporomandibular disorders (TMD) who may suffer from clinical problems in the masticatory muscles, the temporomandibular joint and other associated structures.

Millions of people worldwide use their smartphone devices excessively. Prevalence of smartphone addiction among Egyptian university students was 62.4% revealing that females had a higher addiction than men. This excessive use where subjects downwardly flex their neck to enable them to look at the screen, affects head and neck postures leading to forward head posture (FHP) which consequently alters the position of the mandible along with its functions, resulting in an increase tension in the masticatory muscles causing TMD. Addicted smartphone users contribute to changes in craniocervical region which led to myogenic TMD in young teenagers.

Pain, tenderness in masticatory muscles and cervical muscle endurance are common clinical findings in patients with TMD; where muscle tenderness is reduced and cervical muscle endurance was found to have a shorter duration holding time when performing neck extensor endurance test due to higher fatigability of neck extensor muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age range from 18 - 40 years.
2. Both males and females will be recruited.
3. Subjects diagnosed as myogenic TMD according to the presence of trigger points in masseter, temporalis, upper trapezius and C5-C6 articular pillars according to the myofascial diagnostic criteria that includes a taut band and hypersensitive spot
4. All subjects are heavy smartphones users, using the SAS-SV, the cuffof value for males is 31 and for females is 33.
5. All subjects will have forward head posture assessed by CVA less than 49.9 degrees.

Exclusion Criteria:

1. History of head, neck or TMJ trauma
2. Patients who underwent orthodontic treatment
3. Congenital, or acquired postural deformity
4. No previous neck or spinal or TMJ surgery
5. Subjects who are on anti-inflammatory or analgesic drugs for pain

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 23 subjects with myogenic TMD, FHP and addicted to smartphone devices will be assessed for pressure pain threshold on trigger points and muscle endurance in both masticatory and neck muscles
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | 5 mintues
  For the masticatory muscles, the subject will be sitting and the therapist will place the pressure algometer on the belly of the masseter and temporalis muscles. A gradual pressure will be applied until the subject experiences pain. The value displayed on the device will be recorded. This will be repeated 3 times on each side. For the upper trapezius muscles, subject will be seated. Using the algometer, a pressure will be applied on midpoint of the trapezius. Then subject will lie prone, to apply pressure by the algometer on a point 1 cm laterally to the midpoint between C6 and C5 spinous processes. A value will be recorded when subject feels pain. This will be repeated 3 times on each side.

SECONDARY OUTCOMES:
muscle endurance | 10 minutes
  To assess masticatory muscles, subject will sit in an upright position and will bite on the first molar at maximum voluntary contraction until exhaustion on an I load mini bite load cell. Using a stopwatch, time in seconds will be recorded for both sides. long maintenance time means good endurance.Test will be terminated when any pain or discomfort is felt in the masticatory muscles.Craniocervical extension endurance test will assess neck extensors endurance. Subject will lie prone on a plinth with the head and neck unsupported and a bubble inclinometer will be fixed on the head using a strap. Subject will be asked to sustain a neutral position for as long as possible and time in seconds will be recorded. The test will be terminated if pain is felt in the neck or if the head failed to maintain its neutral position or if it moved more than 5 degrees shown by inclinometer.
smartphone addiction scale short version | 2 minutes
  Smartphone addiction scale - short version (SAS-SV) is a screening tool to identify individuals that are dependent on smartphone use. Maximum score is 60 and the minimum is 10. The cut off value of smartphone addiction use differ by gender, in males it is 31 and in females it is 33. higher score means patient were addicted on the smartphones.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Egyptian University, Cairo, Egypt

REFERENCES:
- [Background] Resende CM, Alves AC, Coelho LT, Alchieri JC, Roncalli AG, Barbosa GA. Quality of life and general health in patients with temporomandibular disorders. Braz Oral Res. 2013 Mar-Apr;27(2):116-21. doi: 10.1590/s1806-83242013005000006. Epub 2013 Mar 1. PMID 23459771
- [Background] Rashed, S. A., & Elsharkawy, A. T. (2018). Prevalence and severity of Temporomandibular disorders signs and symptoms Among Students of The Ahram Canadian University (ACU). Egyptian Dental Journal, 64(3-July (Oral Surgery), 2097-2104
- [Background] Soliman Elserty, N., Ahmed Helmy, N., & Mohmed Mounir, K. (2020). Smartphone addiction and its relation to musculoskeletal pain in Egyptian physical therapy students. European Journal of Physiotherapy, 22(2), 70-78
- [Background] Kee IK, Byun JS, Jung JK, Choi JK. The presence of altered craniocervical posture and mobility in smartphone-addicted teenagers with temporomandibular disorders. J Phys Ther Sci. 2016 Jan;28(2):339-46. doi: 10.1589/jpts.28.339. Epub 2016 Feb 29. PMID 27065516
- [Background] Berolo S, Wells RP, Amick BC 3rd. Musculoskeletal symptoms among mobile hand-held device users and their relationship to device use: A preliminary study in a Canadian university population. Appl Ergon. 2011 Jan;42(2):371-8. doi: 10.1016/j.apergo.2010.08.010. Epub 2010 Sep 15. PMID 20833387
- [Background] Mani, M. S., Ahamed, S. Y., Kavithagiri, N. L., Ambiga, P., Sivaraman, G., & Balan, N. (2019). Association of Mobile Phone Usage in Patients with Temporomandibular Joint Disorders-A Comparative Study. Journal homepage: www. nacd. in Indian J Dent Adv, 11(3), 79-85.
- [Background] Park, J., Kim, K., Kim, N., Choi, I., Lee, S., Tak, S., & Yim, J. (2015)b. A comparison of cervical flexion, pain, and clinical depression in frequency of smartphone use. International Journal of Bio-Science and Bio-Technology, 7(3), 183-90
- [Background] Torkamani MH, Mokhtarinia HR, Vahedi M, Gabel CP. Relationships between cervical sagittal posture, muscle endurance, joint position sense, range of motion and level of smartphone addiction. BMC Musculoskelet Disord. 2023 Jan 23;24(1):61. doi: 10.1186/s12891-023-06168-5. PMID 36690958
- [Background] Vargas CM, Kramarow EA, Yellowitz JA. The oral health of older Americans. Aging Trends. 2001 Mar;(3):1-8. No abstract available. PMID 11894225
- [Background] Hugo FN, Hilgert JB, de Sousa Mda L, da Silva DD, Pucca GA Jr. Correlates of partial tooth loss and edentulism in the Brazilian elderly. Community Dent Oral Epidemiol. 2007 Jun;35(3):224-32. doi: 10.1111/j.0301-5661.2007.00346.x. PMID 17518969
- [Background] Svensson P, Macaluso GM, De Laat A, Wang K. Effects of local and remote muscle pain on human jaw reflexes evoked by fast stretches at different clenching levels. Exp Brain Res. 2001 Aug;139(4):495-502. doi: 10.1007/s002210100806. PMID 11534874
- [Background] Martinez-Merinero P, Nunez-Nagy S, Achalandabaso-Ochoa A, Fernandez-Matias R, Pecos-Martin D, Gallego-Izquierdo T. Relationship between Forward Head Posture and Tissue Mechanosensitivity: A Cross-Sectional Study. J Clin Med. 2020 Feb 27;9(3):634. doi: 10.3390/jcm9030634. PMID 32120895
- [Background] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462
- [Background] Diab AA, Moustafa IM. The efficacy of forward head correction on nerve root function and pain in cervical spondylotic radiculopathy: a randomized trial. Clin Rehabil. 2012 Apr;26(4):351-61. doi: 10.1177/0269215511419536. Epub 2011 Sep 21. PMID 21937526
- [Background] Yao Y, Cai B, Xu LL, Wang JW. [Correlation between neck pressure pain threshold and forward head posture in patients with temporomandibular joint disorders]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2021 Aug 9;56(8):759-763. doi: 10.3760/cma.j.cn112144-20210312-00111. Online ahead of print. Chinese. PMID 34404141